CLINICAL TRIAL: NCT06660004
Title: The Effects of 8-Week Creatine HCl and Creatine Ethyl Ester Supplementation on Cognitive Performance, Multidimensional Fatigue, Brain Metabolism, and Biochemical Indices in Perimenopausal and Menopausal Women
Brief Title: Creatine HCl and Creatine Ethyl Ester Supplementation in Perimenopausal and Menopausal Women
Acronym: CONCRET-MENOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, Head of the Applied Bioenergetics Lab, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CC-1-24
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Menopausal; Perimenopause
Keywords: creatine; brain metabolism; cognition; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Creatine hcl (Experimental): One capsule per day of creatine hcl during breakfast
  Interventions: Dietary Supplement: Dietary Supplement: Experimental 1 Creatine HCl
- Creatine hcl 2 (Experimental): One capsule during breakfast and one during dinner of creatine hcl
  Interventions: Dietary Supplement: Dietary Supplement: Experimental 2 Creatine HCl
- Creatine ethyl ester (Experimental): One capsule during breakfast and one during dinner of creatine ethyl ester
  Interventions: Dietary Supplement: Dietary Supplement: Experimental 3 Creatine Ethyl ester
- Placebo (Placebo Comparator): One capsule per day of inulin during breakfast
  Interventions: Dietary Supplement: Dietary Supplement: Experimental 4 Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Experimental 1 Creatine HCl — Creatine hcl
  Arms: Creatine hcl
Dietary Supplement: Dietary Supplement: Experimental 2 Creatine HCl — Creatine hcl
  Arms: Creatine hcl 2
Dietary Supplement: Dietary Supplement: Experimental 3 Creatine Ethyl ester — Creatine ethyl ester
  Arms: Creatine ethyl ester
Dietary Supplement: Dietary Supplement: Experimental 4 Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled double-blind parallel-group interventional trial is to evaluate the effects of of dietary supplementation with creatine HCl and creatine ethyl ester supplementation on cognitive performance, multidimensional fatigue, brain metabolism, and biochemical indices in perimenopausal and menopausal women

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5 - 29.9 kg/m2
* Free of major chronic diseases or acute disorders (including AD and dementia (MMSE score > 25 points)
* MENOPAUSAL: no menstrual cycle for consecutive 12 months (with no other obvious causes)
* PERIMENOPAUSAL: Still menstruating (regular or irregular) but have at least one of the following symptoms: (1) hot flashes, (2) sleep disturbances, (3) mood swings, and (4) concentration difficulties
* Given written informed consent

Exclusion Criteria:

* History of dietary supplement use 4 weeks before the study commences
* Pregnancy (or planning pregnancy)
* Abnormal values for lab clinical chemistry (> 2 SD)
* Unwillingness to return for follow-up analysis
* Participation in other clinical trials

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Fatigue | Change from baseline fatigue at 8 weeks
  Level of fatigue as assessed by the Multidimensional Fatigue Inventory (MFI)

SECONDARY OUTCOMES:
Time to exhaustion | Change from baseline time to exhaustion at 8 weeks
  Running time to exhaustion during incrementaltestontreadmill
Brain creatine | Change from baseline brain creatine concentrations at 8 weeks
  Magnetic resonance spectra for brain creatine concentrations
Cognitive interference | Change from baseline fatigue at 8 weeks
  Ability to inhibit cognitive interference as assessed by the The Stroop Color and Word Test
Amyloid b | Change from baseline time to exhaustion at 8 weeks
  Serum levels of amyloid b

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — Applied BIoenergetics Lab
Locations (1):
- FSPE Applied BIoenergetcis Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in perimenopause. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in perimenopause.
URL: https://www.appliedbioenergetics.org/

REFERENCES:
- [Background] Ostojic SM, Stea TH, Ellery SJ, Smith-Ryan AE. Association between dietary intake of creatine and female reproductive health: Evidence from NHANES 2017-2020. Food Sci Nutr. 2024 Apr 30;12(7):4893-4898. doi: 10.1002/fsn3.4135. eCollection 2024 Jul. PMID 39055234
- [Derived] Korovljev D, Ostojic J, Panic J, Ranisavljev M, Todorovic N, Nedeljkovic D, Kuzmanovic J, Vranes M, Stajer V, Ostojic SM. The Effects of 8-Week Creatine Hydrochloride and Creatine Ethyl Ester Supplementation on Cognition, Clinical Outcomes, and Brain Creatine Levels in Perimenopausal and Menopausal Women (CONCRET-MENOPA): A Randomized Controlled Trial. J Am Nutr Assoc. 2025 Aug 25:1-12. doi: 10.1080/27697061.2025.2551184. Online ahead of print. PMID 40854087